CLINICAL TRIAL: NCT07186348
Title: Efficacy of Ice Packing Application in Post-Hemorrhoidectomy Recovery: A Propensity Score-Matched Study
Brief Title: Efficacy of Ice Packing Application in Post-Hemorrhoidectomy Recovery
Acronym: ICE-HEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301650B0
Record Dates: First submitted 2025-06-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Hemorrhoids Third Degree; Hemorrhoids Fourth Degree; Hemorrhoids
Keywords: Ice packing; Cryotherapy; Hemorrhoidectomy; Postoperative pain; Acute urine retention
MeSH Terms: conditions — Pain, Postoperative; Hemorrhoids | interventions — Cryotherapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice packing Group (Active Comparator): Ice packing with standard care
  Interventions: Procedure: Ice packing; Procedure: Standard Care (in control arm)
- Standard care group (Active Comparator): Standard care
  Interventions: Procedure: Standard Care (in control arm)

INTERVENTIONS:
Procedure: Ice packing — 10 minutes ice packing application after surgery
  Other Names: Cryotherapy
  Arms: Ice packing Group
Procedure: Standard Care (in control arm) — Standard Care (in control arm)

SUMMARY:
According to the previous study, surgical intervention exhibited significant differences in daily life before and after a hemorrhoidectomy. However, post-hemorrhoidectomy pain remains a challenging problem, and the incidence of moderate to severe post-hemorrhoidectomy pain could be as high as 65%. In particular, post-hemorrhoidectomy pain management remains unsolved in 5% of cases who remains severe pain despite standard pain management which potentially leads to a longer hospital stay and more opioid requirement.

Post-hemorrhoidectomy pain arises from multiple pathological mechanisms. Tissue trauma during the surgical procedure activates nociceptors in the richly innervated anal region. The subsequent inflammatory response releases cytokines, leading to localized edema and increased nerve sensitivity. Anal sphincter spasm, a common postoperative response, further exacerbates pain by creating tension around the surgical site. Additionally, defecation can mechanically irritate the wound, particularly in cases of hard stools or straining, further aggravating discomfort.

The benefits of cold therapy have been recognized for thousands of years. By lowering tissue temperature through ice packing, it is believed that blood flow, pain, metabolism, and muscle spasms can be reduced, thereby minimizing inflammation and promoting the recovery of soft-tissue injuries. Ice therapy has been shown to be a safe and effective method for postoperative pain management in various procedures, including orthopedic surgery, maxillofacial surgery, laparotomy and laparoscopic surgery, thoracic surgery, hernia repair, and gynecologic of postpartum care.

Our study hypothesized that the postoperative ice packing application in hemorrhoidectomy patients could help to manage post-hemorrhoidectomy pain, leading to either reduced narcotic consumption or improved pain control compared to patients who did not use ice packing application, and while ensuring patients' safety during the surgical intervention. The study aimed to assess the effectiveness of ice packing application versus the standard of care in relieving pain following hemorrhoidectomies.

DETAILED DESCRIPTION:
Data were collected from patients diagnosed with grade III or IV hemorrhoids who underwent surgical intervention between January 2021 and September 2022 at the Keelung branch of Chang Gung Memorial Hospital, Taiwan. Clinical demographic data, medication history, hemorrhoid-related characteristics, operative details, postoperative pain scores, and outcomes were retrieved from the hospital's electronic medical records. Patient demographics and medication histories-including age, gender, American Society of Anesthesiologists (ASA) classification, Eastern Cooperative Oncology Group (ECOG) performance status, body mass index (BMI), tobacco use, and comorbidities-were recorded. Hemorrhoid-related characteristics, such as symptoms, disease grading, and the number of hemorrhoidectomy quadrants, were also documented. Operative characteristics and postoperative outcomes were recorded, including length of hospital stay, number of outpatient department (OPD) visits, operative time and surgical devices used, complications, painkiller usage, and postoperative Numeric Rating Scale (NRS) pain score. Postoperative complications included acute urinary retention (AUR), bleeding, stool impaction, prolonged hospital stay, and readmission rates were also recorded. All patients were followed until September 2023 or until follow-up visits were no longer required. The median follow-up period was 2 months. All data collection and analysis procedures were approved by the Institutional Review Board of Chang Gung Memorial Hospital, Taiwan (IRB No. 202301650B0).

This retrospective cohort study initially included 480 consecutive patients with grade III or IV hemorrhoids who underwent surgical intervention. Patients who also underwent additional anorectal surgeries-such as fistulectomy (n=16), ulcerectomy (n=14), isolated external skin tag excision (n=3)-or had incomplete data (n=18) were excluded, leaving 429 patients eligible for inclusion. Ice packing was introduced and application starting in August 2021. Based on the surgery date, patients were divided into two groups: the standard care group (before August 2021) and the ice packing group (after August 2021). To address selection bias inherent to this non-randomized study and achieve balanced covariates across the groups, propensity score matching (PSM) was performed using a logistic regression model, with the use of ice packing as the dependent variable. Patients in both groups were matched based on clinical characteristics, including sex, age, ASA, BMI, smoking status, comorbidities, disease grading, number of hemorrhoidectomy quadrants, surgical device, and postoperative pain management. A 1:1 PSM was conducted using the nearest neighbor matching method with a caliper width of 0.2.

All patients underwent standard preoperative preparation and pre-anesthesia evaluation. Surgical procedures were performed by five experienced surgeons, with the operation's extent determined by hemorrhoid grading. LigaSure™, a single-use, self-funded energy device, was used with patient consent. Patients taking anticoagulants (e.g., Clopidogrel, apixaban, dabigatran, edoxaban, rivaroxaban, and warfarin) were instructed to discontinue their medications 5 to 7 days before surgery and resume them 24 to 48 hours post-surgery. Antiplatelet agents, such as aspirin, were continued during the perioperative period.

The surgical procedure was as follows: patients were positioned in the Sims position under mask-induced general anesthesia. A digital examination and anoscopy were performed, followed by an injection of lidocaine and adrenaline (10,000:1) to provide additional local anesthesia and facilitate mucosal dissection. Hemorrhoid complexes requiring excision were clearly identified. The Ferguson procedure was then performed. For patients opting for LigaSure™-assisted hemorrhoidectomy, excision and dissection followed the same protocol using the device. After achieving adequate hemostasis, the apex of each hemorrhoid pedicle was suture-ligated, and the mucosal and skin wounds were closed with 4-0 Polysorb™ sutures. At the conclusion of the procedure, sebacoyl dinalbuphine ester (SDE), a single-dose, extended-release nalbuphine prodrug, was administered as self-funded analgesia with patient consent. In the ice packing group, a 10-minute ice packing application was performed postoperatively. The ice packing device, featuring a tissue fluid collection plastic test tube and condom, is illustrated in Figure 2, and Figure 3 illustrates the diagram utilized during the surgical procedure.

Post-surgery, intravenous fluids were discontinued upon waking from anesthesia. Patients were prescribed 1000 mg of mefenamic acid with 250 mg of magnesium oxide, taken four times daily. Sitz baths and wound care with neomycin ointment were performed twice daily as part of the routine postoperative care protocol. Morphine (5 mg) was administered via intramuscular injection every 6 hours if wound pain was intolerable. Additionally, parecoxib, a selective cyclooxygenase-2 (COX-2) inhibitor, was offered as self-funded analgesia via intravenous injection every 12 hours with patient consent. Patients were discharged on postoperative days 1 to 3 following smooth urination.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with grade III or IV hemorrhoids who underwent Ferguson hemorrhoidectomy

Exclusion Criteria:

* Patients who also underwent additional anorectal surgeries-such as fistulectomy, ulcerectomy, isolated external skin tag excision
* Patients with incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
NRS pain scores | From day of surgery till postoperative day 2, assessed up to 5 years
  NRS pain scores on the day of surgery and on the first postoperative day using Numeric Rating Scale(0 is equivalent to no pain and 10 indicates the worst possible pain)

SECONDARY OUTCOMES:
Acute urine retention | From day of surgery till postoperative day 2, assessed up to 5 years
  The sudden inability to void, usually associated with bloating, severe urgency, general distress, lower abdominal distension, and suprapubic pain
Postoperative bleeding | From day of surgery up to 1 month, assessed up to 5 years
  Bleeding occurring after completion of a surgical procedure, which may occur immediately or may be delayed, and which may or may not be wound related
Prolonged hospital stay | From day of surgery up to day of discharge, assessed up to 5 years
  A hospital admission that lasts longer than what is considered typical or expected for a particular condition or procedure. In patients particularly post-hemorrhoidectomy, 3 days admission is expected.
Opioids consumption | From day of surgery till day of discharge, assessed up to 5 years
  Opioids consumption in administration frequency(n) and total doses(mg) needed for pain control post-hemorrhoidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Keelung Branch, Keelung, Taiwan, Taiwan